CLINICAL TRIAL: NCT01577966
Title: A Pilot Study to Determine the Effect of Sulfasalazine on Glutamate Levels Detected by Magnetic Resonance Spectroscopy(MRS) in Patients With Glioma
Brief Title: Pilot Study Effect of Sulfasalazine on Glutamate Levels by(Magnetic Resonance Spectroscopy)MRS in Patients With Glioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Louis Burt Nabors, MD, Professor, Neurology Chair Office, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UAB 1108
Record Dates: First submitted 2012-04-11; First posted 2012-04-16 (Estimated); Results first posted 2016-12-08 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-07

CONDITIONS: Brain Tumor
Keywords: Patients with brain tumors associated with seizures
MeSH Terms: conditions — Brain Neoplasms | interventions — Sulfasalazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sulfasalazine (Experimental)
  Interventions: Drug: Sulfasalazine

INTERVENTIONS:
Drug: Sulfasalazine — Sulfasalazine has been the parent aminosalicylate in use for over 40 years in the treatment of inflammatory bowel disease. The drug is a conjugate of sulfapyridine linked to 5-aminosalicylic acid. In inflammatory bowel disease, the 5-ASA component is the active moiety
  Sulfasalazine is a prodrug that consists of sulfapyridine bonded to mesalamine (5-ASA). Sulfasalazine is cleaved by colonic bacterial azo-reductases into sulfapyridine and the 5-ASA moiety. 5-ASA is metabolized to N-acetyl-5-ASA by an enzyme in the intestinal epithelium and the liver and then excreted in the urine as a mixture of free 5ASA and N-acetyl-5-ASA.

SUMMARY:
The main purpose of this part of the study is to determine the Central Nervous System bioavailability of sulfasalazine.

DETAILED DESCRIPTION:
This is a pilot, open-label, non-randomized, study to determine the effect that orally administered sulfasalazine has on glutamate levels as measured by MRS and on epileptiform spiking as measured by simultaneous MEG/EEG. The intent of the dose escalation is to determine an Optimal Biological Dose (OBD) based on changes in tumor glutamate levels. The OBD is defined as the dose that has the maximal reduction in tumor glutamate levels after normalization to uninvolved brain.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be > 18 years of age or older.
2. Patients must have histologically proven low grade astrocytoma,anaplastic astrocytoma, anaplastic mixed glioma, anaplastic oligodendroglioma,glioblastoma multiforme, astrocytoma WHO II,oligodendroglioma WHO II or mixed glioma WHO II. Patients do not haveto demonstrate progressive disease to participate in this study.
3. Patients must have completed initial glioma therapy involving radiation and be 3 months from the completion of radiation therapy. If initial glioma therapy did not include radiation (example: anaplastic oligodendroglioma), then 2 cycles of chemotherapy must be completed prior to study entry.
4. Patients must be maintained on a stable corticosteroid regimen for > 5 days prior to entry.
5. Patients must have a Karnofsky performance status > 60% (i.e. the patient must be able to care for himself/herself with occasional help from others).
6. Patients must have adequate hematologic, renal and liver function (i.e. Absolute neutrophil count > 1500/mm3, Platelets > 100,000/mm3, creatinine > 1.5 mg/dl.
7. Women of childbearing potential must have a negative pregnancy test.
8. Patients with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods to avoid conception. The effect of the investigational drugs on the developing human fetus is not known, but these drugs are likely to be harmful to the developing fetus or nursing infant. Women of child-bearing potential must agree to use adequate contraception (either surgical sterilization; approved hormonal contraceptives such as birth control pills: Depo-Provera, or Lupron Depot; barrier methods such as condom or diaphragm along with spermicide; or an IUD). Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician and study PI immediately.
9. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Pregnant or breast feeding.
2. Exclude sexually active males and females unwilling to practice contraception during the study.
3. Serious concurrent infections.
4. Clinically significant cardiac disease not well controlled with medication (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias) or myocardial infarction within the last 12 months.
5. Patients with other serious uncontrolled co-morbid diseases that the investigator feels may comprise the study findings.
6. Allergic or sensitivity to sulfa containing medications.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis B Nabors, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sulfasalazine: Sulfasalazine
Period: Overall Study
Arm/Group | Sulfasalazine
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sulfasalazine
Number analyzed (Participants) | 9
Age, Continuous [Mean (Full Range); unit: years] | 43 [25 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Percent Decrease in Central Nervous System Bioavailability of Sulfasalazine
Description: To determine the ability of sulfasalazine to alter glioma glutamate levels. These levels will be measured by Magnetic Resonance Spectroscopy (MRS). The percent change is noted per subject. The measure is a % decrease of glioma glutamate levels
Time Frame: up to 2 years post baseline
Measure: Number; unit: percentage of change
Arm/Group | Sulfasalazine
Number analyzed (Participants) | 9
percentage of change
  GBM Pt 2 | 17
  GBM Pt 1 | 23
  GBM Pt 4 | 28
  Astro Pt 3 | 5
  Astro Pt 9 | 55
  Astro Pt 5 | 58
  Oligo Pt 8 | 12
  Oligo Pt 6 | 18
  Oligo Pt 7 | 42

ADVERSE EVENTS:
Time Frame: AEs and SAEs were not collected or recorded for these subjects.
Arm/Group | Sulfasalazine
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No